CLINICAL TRIAL: NCT05508243
Title: Dermatologist-supervised Assessment of Primary and Accumulated Irritation Potential and Skin Sensitization Potential for the NASAL SPRAY Product
Brief Title: Dermatological Assessment of Primary Dermal Irritability Accumulated and Sensitization of Hyaluronic Nasal Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HB053-22
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Sensitivity, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Hyaluronic Nasal Spray

INTERVENTIONS:
Other: Hyaluronic Nasal Spray — Health care product - nasal application

SUMMARY:
Evaluate the potential of Primary Dermal Irritability, Accumulated Dermal Irritability and Dermal Sensitization, of health products through the application of Patch Test, proving the safety of the product for topical use. The study will be conducted with a Brazilian sample in which 65 research participants will be included. Depending on the results, the present study may support the claim: dermatologically tested.

ELIGIBILITY:
Inclusion Criteria:

* Healthy research participant
* Age range between 18 and 70 years.
* Gender: female and male.
* Phototype (Fitzpatrick): I to IV.
* Agree to adhere to the requirements of the study in the fight against the COVID-19 pandemic, through preventive measures: use a mask according to WHO guidelines; use the mask while traveling to the research center and during the study procedures; maintain social distancing; wash hands frequently with soap and/or alcohol gel and go to the research center only at scheduled times to avoid agglomerations.
* Agree not to wet the site during the entire test period;
* Understand the test procedures and agree to their adherence to the study requirements;
* Absence of inflammatory dermatoses or tattoo at the application site;
* Signing of the Free and Informed Consent Term (FICT).

Exclusion Criteria:

* Pregnancy, lactation;
* Participants with hyperthermia (body temperature greater than or equal to 37.5ºC);
* Participants who have been diagnosed with COVID-19 by RT-PCR exam or by the presence of IgM antibodies in the serology exam, in the last 4 weeks or who are presenting the following symptoms: dry or productive cough, sneezing, runny nose, body pain , headache, anosmia (loss of smell), ageusia (loss of taste) and/or any other symptom that may be related to covid-19 at the discretion of the investigator;
* Participant who belongs to the risk group for COVID-19, that is, with cardiovascular, renal and chronic respiratory problems, immunosuppressed or other conditions that the doctor judges as belonging to the risk group;
* Participants with heart disease (eg, but not limited to: atrial fibrillation, obstructive coronary artery disease);
* Participants with renal and/or neurological diseases;
* Participants with severe or decompensated lung and/or respiratory diseases;
* Use of corticosteroids, antihistamines and/or anti-inflammatory drugs;
* Presence of localized or generalized skin diseases;
* Presence of active inflammatory dermatoses in the test region;
* Frequent exposure to the sun or tanning beds;
* Have participated in an allergenicity study within a period of less than four weeks from the beginning of the study;
* Research participants with a history of allergy to the material used in the study;
* Atopy history;
* History of pathologies aggravated or triggered by ultraviolet radiation;
* Immunodeficiency carriers;
* Forecast of intense sun exposure or tanning session during the study period;
* Forecast to take a bath in the sea, swimming pool or sauna during the study;
* Research participants who practice water sports;
* Research participants with dermographism;
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-steroidal anti-inflammatory drugs, and corticosteroids up to 2 weeks before selection;
* Treatment with acidic vitamin A and/or its derivatives orally or topically up to 1 month before the start of the study;
* Aesthetic and/or dermatological body treatment up to 03 weeks before selection;
* Vaccination forecast during the study or up to 03 weeks before the study;
* Any condition not mentioned above that, in the opinion of the investigator, could compromise the evaluation of the study;
* History of non-adherence or unwillingness to adhere to the study protocol;
* Professionals directly involved in carrying out this protocol and their families.
* Be participating in some other study at the moment.
* Any condition that, in the opinion of the researcher, could compromise the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Absence | 6 weeks
  Absence occurence of phototoxicity and photoallergy

CONTACTS AND LOCATIONS:
Locations (1):
- Kosmoscience Ciência e Tecnologia Cosmética Ltda, Campinas, São Paulo, Brazil